CLINICAL TRIAL: NCT00907738
Title: A Continuation Clinical Trial of Oral Vorinostat (MK-0683) in Advanced Cancers
Brief Title: A Continuation Clinical Trial of Oral Vorinostat (MK-0683) in Advanced Cancers (MK-0683-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-007; 2009_595; NCT00588055 (obsolete NCT alias)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat (Experimental)
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — All patients will receive vorinostat at the same dose and schedule as they received in the base protocol until disease progression or unacceptable toxicity.
  Other Names: MK-0683

SUMMARY:
This study will evaluate the safety and tolerability of continuing vorinostat (MK-0683) dosing in cancer patients previously enrolled in one of five base studies (MK-0683-001, MK-0683-006, MK-0683-008, MK-0683-012, or MK-0683-013) who have shown benefit from receiving this drug.

ELIGIBILITY:
Inclusion Criteria:

* Patient participated in one of the five vorinostat base protocols, has not shown tumor progression on that study, and has tolerated the study drug
* Patient did not withdraw from the base protocol
* Patient agrees to practice effective birth control during the study

Exclusion Criteria:

* Patient is receiving other standard and/or investigational anticancer therapy
* Patient has any condition or disease that would interfere with compliance or pose addition risk in administering the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Duvic M, Olsen EA, Breneman D, Pacheco TR, Parker S, Vonderheid EC, Abuav R, Ricker JL, Rizvi S, Chen C, Boileau K, Gunchenko A, Sanz-Rodriguez C, Geskin LJ. Evaluation of the long-term tolerability and clinical benefit of vorinostat in patients with advanced cutaneous T-cell lymphoma. Clin Lymphoma Myeloma. 2009 Dec;9(6):412-6. doi: 10.3816/CLM.2009.n.082. PMID 19951879

RESULTS

PARTICIPANT FLOW:
Groups:
- Base Protocol 001: Vorinostat 400 mg daily (QD)
- Base Protocol 006: vorinostat 200 mg twice daily (BID)
- Base Protocol 008: vorinostat 400 mg QD
- Base Protocol 012: 400 mg QD 7/21 (7 days of dosing followed by 14 days rest every 21 day cycle) + pemetrexel & cisplatin OR 300 mg BID 3/7 (3 days of dosing followed by 7 days rest every first week followed by 2 weeks off) OR 300 mg QD 14/21 (14 days of dosing followed by 7 days rest every 21 day cycle) OR 300 mg QD 7/21 (7 days of dosing followed by 14 days rest every 21 day cycle) + pemetrexel
- Base Protocol 013: vorinostat 200 mg BID 14/21 OR 300 mg BID 3/7 (3 days dosing followed by 4 days rest every week)
Period: Overall Study
Arm/Group | Base Protocol 001 | Base Protocol 006 | Base Protocol 008 | Base Protocol 012 | Base Protocol 013
Started | 13 | 1 | 7 | 4 | 2
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 1 | 7 | 4 | 2
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0
Not completed — not specified or withdrew consent | 3 | 0 | 0 | 0 | 0
Not completed — Disease progression | 8 | 1 | 6 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Protocol 001 | Base Protocol 006 | Base Protocol 008 | Base Protocol 012 | Base Protocol 013 | Total
Number analyzed (Participants) | 13 | 1 | 7 | 4 | 2 | 27
Age, Customized [Number; unit: Participants] — All participants were at least 18 years of age.
  Participants | 13 | 1 | 7 | 4 | 2 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 4 | 1 | 2 | 15
  Male | 5 | 1 | 3 | 3 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Serious Drug-related Adverse Event (AE)
Description: A serious adverse event (SAE) was any AE occurring at any dose that resulted in death, was life-threatening, resulted in a persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, or was an overdose.
  A drug-related SAE was one that was thought to be possibly, probably, or definitely related to the study drug.
Time Frame: From the first dose of study drug until the patient experiences disease progression, withdraws consent, or develops unacceptable toxicity (from Day 1 up to 4 years and 9 months)
Measure: Number; unit: percent of participants
Arm/Group | Base Protocol 001 | Base Protocol 006 | Base Protocol 008 | Base Protocol 012 | Base Protocol 013
Number analyzed (Participants) | 13 | 1 | 7 | 4 | 2
percent of participants | 7.7 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The MedDRA version used for protocol 001 was 13.0 For all the other protocols (006, 008,012, and 013), the MedDRA version used was 11.1.
  Non-serious adverse events were only collected if they caused drug interruption, discontinuation, or dose reduction.
Arm/Group | Base Protocol 001 (Vorinostat 400 mg Once Daily [QD]) | Base Protocol 006 (Vorinostat 200 mg Twice Daily [BID]) | Base Protocol 008 (Vorinostat 400 mg Once Daily [QD]) | Base Protocol 012 (Vorinostat 400 mg Once Daily [QD] 7/21) | Base Protocol 012 (Vorinostat 300 mg Twice Daily [BID] 3/7) | Base Protocol 012 (Vorinostat 300 mg Once Daily [QD] 14/21) | Base Protocol 012 (Vorinostat 300 mg Once Daily [QD] 7/21) | Base Protocol 013 (Vorinostat 200 mg Twice Daily [BID] 14/21) | Base Protocol 013 (Vorinostat 300 mg Twice Daily [BID] 3/7)
Serious Adverse Events (participants affected / at risk) | 4/13 | 1/1 | 1/7 | 0/1 | 1/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 6/13 | 0/1 | 2/7 | 0/1 | 1/1 | 0/1 | 0/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Protocol 001 (Vorinostat 400 mg Once Daily [QD]) (N=13) | Base Protocol 006 (Vorinostat 200 mg Twice Daily [BID]) (N=1) | Base Protocol 008 (Vorinostat 400 mg Once Daily [QD]) (N=7) | Base Protocol 012 (Vorinostat 400 mg Once Daily [QD] 7/21) (N=1) | Base Protocol 012 (Vorinostat 300 mg Twice Daily [BID] 3/7) (N=1) | Base Protocol 012 (Vorinostat 300 mg Once Daily [QD] 14/21) (N=1) | Base Protocol 012 (Vorinostat 300 mg Once Daily [QD] 7/21) (N=1) | Base Protocol 013 (Vorinostat 200 mg Twice Daily [BID] 14/21) (N=1) | Base Protocol 013 (Vorinostat 300 mg Twice Daily [BID] 3/7) (N=1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Protocol 001 (Vorinostat 400 mg Once Daily [QD]) (N=13) | Base Protocol 006 (Vorinostat 200 mg Twice Daily [BID]) (N=1) | Base Protocol 008 (Vorinostat 400 mg Once Daily [QD]) (N=7) | Base Protocol 012 (Vorinostat 400 mg Once Daily [QD] 7/21) (N=1) | Base Protocol 012 (Vorinostat 300 mg Twice Daily [BID] 3/7) (N=1) | Base Protocol 012 (Vorinostat 300 mg Once Daily [QD] 14/21) (N=1) | Base Protocol 012 (Vorinostat 300 mg Once Daily [QD] 7/21) (N=1) | Base Protocol 013 (Vorinostat 200 mg Twice Daily [BID] 14/21) (N=1) | Base Protocol 013 (Vorinostat 300 mg Twice Daily [BID] 3/7) (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Non-serious adverse events were only collected if they caused drug interruption, discontinuation, or dose reduction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.